CLINICAL TRIAL: NCT00000370
Title: Treatment of Social Phobia: Mediators And Moderators
Brief Title: Treatment of Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stefan G. Hofmann, Professor of Psychology, Boston University Charles River Campus
Purpose: Treatment
Other Study IDs: R29MH057326 (NIH); R29MH057326 (NIH); DSIR AT-AS
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Phobic Disorders; Social Phobia; Public Speaking Anxiety
Keywords: Cognitive Therapy; Cost of Illness; Female; Human; Male; Phobic Disorders; Phobic Disorders -- *therapy; Phobic Disorders -- pathology
MeSH Terms: conditions — Phobic Disorders; Phobia, Social | interventions — Cognitive Behavioral Therapy; Psychosocial Intervention

INTERVENTIONS:
Behavioral: Cognitive behavior therapy
Behavioral: Performance-based exposure therapy
Behavioral: Psychosocial intervention

SUMMARY:
Social phobia is a very common and debilitating disorder, with public speaking anxiety being the most common fear. Psychologists have found that treating patients for their fear of public speaking, through cognitive-behavioral treatment (talk-based therapy) or exposure treatment (where participants participate in actual public speaking sessions), not only helps patients overcome this fear but also helps them overcome their more general social fears. However, little is known about how this change occurs during therapy. This study tries to identify the factors that contribute most to successful therapy.

Patients are assigned randomly (like tossing a coin) to 1 of 3 groups. Group 1 will receive cognitive-behavioral treatment and Group 2 will receive exposure treatment. Group 3 will not receive treatment. Study leaders will monitor patient response to treatment through behavioral tests and assessments.

An individual may be eligible for this study if he/she:

Has social phobia with public speaking anxiety.

DETAILED DESCRIPTION:
The primary goal of the present study is to identify the mediators and moderators of change in the treatment of social phobia and, in so doing suggest a common mechanism of action for all brief psychosocial interventions. Perceived self-efficacy of social behavior, negative cognitive appraisal (estimated social costs), and perceived emotional control will be considered as potential mediators; avoidant personality disorder and the generalized subtype of social phobia will be considered as potential predictors for poor treatment outcome.

Social phobia is a very prevalent and debilitating disorder, with public speaking anxiety being the most common fear among socially phobic individuals. Although there are a number of effective psychosocial treatments for social phobia (e.g., cognitive-behavioral treatments and exposure therapy) very little is known about the underlying mechanism of therapeutic change (i.e., the mediators of change), and the variables that are predictive of treatment outcome (i.e., the moderators of change). Furthermore, it is unclear why treating individuals for their public speaking anxiety can generalize to other untreated social fears.

Patients are randomly assigned to either a comprehensive cognitive-behavioral treatment for social phobia (n=43), a performance-based exposure treatment for public speaking anxiety without cognitive intervention (n=43), or a waitlist control group (n=43). Clinician ratings, behavioral tests, cognitive assessments, subjective ratings, and physiological measures are employed to determine the degree of therapeutic gains in various social phobia domains. The main hypothesis is that perceived emotional control will mediate treatment outcome and generality of effectiveness independent of the specific treatment condition.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Social phobia with public speaking anxiety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-05; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hofmann, PhD, Principal Investigator
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States